CLINICAL TRIAL: NCT04841811
Title: Effectiveness and Safety of Dynamic MRD Guiding Treatment After Aumolertinib Induction Therapy of EGFR-mutation-positive Unresectable Stage III Non-Small Cell Lung Cancer in the MDT Diagnostic Model: an Open-label, Multicenter, Randomized, Phase III Study
Brief Title: MRD Guiding Treatment After Almonertinib Induction Therapy for EGFRm+ Stage III NSCLC in the MDT Diagnostic Model.
Acronym: APPROACH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2101
Record Dates: First submitted 2021-04-01; First posted 2021-04-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
Keywords: EGFR; NSCLC; ctDNA; MDT
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (almonertinib continuous treatment) (Active Comparator): Subjects will be randomly assigned to groups A and B after radical therapy (surgery or radiothrapy) and will receive 110 mg of almonertinib once a day for 2 years or until disease recurrence or metastasis.
  Interventions: Drug: Almonertinib
- Group B (ctDNA monitoring guided the almonertinib treatment) (Experimental): Subjects will be randomly assigned to group B after radical therapy (surgery or radiothrapy) and will receive almonertinib guided by ctDNA dynamic monitoring (every 3 months test ctDNA once, if it is positive, continue to receive almonertinib 110 mg once a day, if it is negative, stop almonertinib until ctDNA turns positive and receive almonertinib treatment again).
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — ctDNA dynamic monitoring guided the Almonertinib treatment group after redical surgery orradiotherapy
  Other Names: ctDNA dynamic monitoring guided the Almonertinib treatment

SUMMARY:
This is an open-label, multi-center, randomized, phase III study. It is aimed to firstly evaluate the effectiveness and safety of almonertinib induction therapy in EGFR-mutated patients with unresectable stage III non-small cell lung cancer, and to evaluate the effectiveness and safety of dynamic MRD guided maintenance therapy with almonertinib after induction therapy with almonertinib and local therapy (radical surgery or radiotherapy) evaluated by MDT diagnostic model. The study includes a screening period (not more than 28 days after the subject with signed informed consent before first medication), treatment period (including induction therapy with almonertinib\ radical therapy under MDT model\ consolidation therapy with almonertinib) and follow-up period.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, phase III study. It is aimed to firstly evaluate the effectiveness and safety of almonertinib induction therapy in EGFR-mutated patients with unresectable stage III non-small cell lung cancer, and to evaluate the effectiveness and safety of dynamic MRD guided maintenance therapy with almonertinib after induction therapy with almonertinib and local therapy (radical surgery or radiotherapy) evaluated by MDT diagnostic model. The study includes a screening period (not more than 28 days after the subject with signed informed consent before first medication), treatment period (including induction therapy with almonertinib\ radical therapy under MDT model\ consolidation therapy with almonertinib) and follow-up period.

Eligible subjects receive 110 mg of almonertinib once a day for 8 consecutive weeks of induction therapy; local treatment (surgical or radical radiotherapy) is selected after MDT assessment. Subjects will be randomly assigned to groups A and B. Stratification factors included EGFR 19deletion or EGFR 21L858R mutation; shedding or non-shedding ctDNA at baseline; radical surgery or radiotherapy under MDT model.

Subjects in group A will receive 110 mg of almonertinib once a day for 2 years. Imaging evaluation is conducted every 12 weeks. Subjects in group B will receive almonertinib guided by dynamic MRD monitoring. When ctDNA was positive (MRD+), subjects will receive 110 mg of almonertinib once a day for 12 weeks; when ctDNA was negative (MRD-), subjects will stop almonertinib and be observed for 12 weeks. This model will continue until disease recurrence or metastasis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be included in this study:

1. Over 18 years old (including 18 years old) and under 70 years old (including 70 years old).
2. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0 or 1, and there is no deterioration within 2 weeks before the study drug treatment, and the expected survival period is not less than 12 weeks.
3. Stage III non-squamous cell non-small cell lung cancer confirmed by histopathology or cytology and determined by the investigator to be unresectable (International Association for the Study of Lung Cancer Eighth Edition Lung Cancer Staging).
4. Tumor tissue samples or blood samples, pleural effusions, ascites effusions, and pericardial effusions are confirmed to be EGFR sensitive mutations (ie, exon 19 deletion or L858R, alone or coexisting, Or with other EGFR mutations, but patients with EGFR20 exon insertion mutations cannot be included in the group) by laboratory tests approved by the investigator.
5. According to the RECIST1.1 standard, the subject must have at least one imaging measurable lesion. The baseline tumor imaging evaluation was performed within 28 days before the first medication.
6. Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and should not breastfeed. Before starting the administration, the pregnancy test is negative, or meeting one of the following criteria proves that there is no risk of pregnancy:

   1. Postmenopausal is defined as age greater than 50 years，and amenorrhea for at least 12 months after stopping all exogenous hormone replacement therapy.
   2. For women younger than 50 years old, if the amenorrhea is 12 months or more after stopping all exogenous hormone treatments, and the luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference value range, also It can be considered postmenopausal.
   3. Have received irreversible sterilization, including hysterectomy, bilateral ovariectomy or bilateral fallopian tube resection, except for bilateral fallopian tube ligation.
7. Male subjects should use barrier contraception (ie, condoms) from screening to 3 months after the study treatment is stopped.
8. The subjects themselves participated voluntarily and signed a written informed consent form.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be included in this study:

1. Have received any of the following treatments:

   1. Have received lung surgery in the past;
   2. Have used any EGFR tyrosine kinase inhibitor in the past;
   3. Previously received any systemic chemotherapy or immunotherapy for lung cancer;
   4. Receive any lung cancer radiotherapy in the past;
2. The patient has undergone open surgery on other parts except the lungs within 14 days before using the study drug for ≤14 days.
3. In addition to NSCLC, another malignant disease has been diagnosed in the past 5 years (excluding completely resected basal cell carcinoma, bladder carcinoma in situ, and cervical carcinoma in situ).
4. Have used proprietary Chinese medicines with anti-tumor effects in the past. Those who have used proprietary Chinese medicines with anti-tumor effects but have been used for no more than 7 days and have been stopped for 2 weeks or more before the drug treatment in this study can be included in the group.
5. There are serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney disease, left ventricular ejection fraction (LVEF) < 50%, uncontrolled hypertension [that is, it is still greater than or equal to CTCAE level 3 hypertension after drug treatment]); suffering from swallowing dysfunction, active gastrointestinal disease, or other significant effects on the absorption of oral drugs, Disorders of distribution, metabolism, and excretion. Those who have had most gastrectomy operations in the past.
6. Fever and body temperature above 38℃ in the past week, or active infection with clinical significance. Active tuberculosis. Active fungal, bacterial and/or viral infections requiring systemic treatment.
7. Those who have active bleeding, new thrombotic diseases, are taking anticoagulant drugs, or have bleeding tendency;
8. The resting electrocardiogram has major clinically significant abnormalities in rhythm, conduction, or morphology, such as complete left bundle branch block, heart block above Ⅱ degree, clinically significant ventricular arrhythmia or atrial fibrillation, Unstable angina pectoris, congestive heart failure, chronic heart failure grade ≥ 2 by the New York Heart Association (NYHA).
9. Myocardial infarction, coronary artery/peripheral artery bypass or cerebrovascular accident occurred within 3 months.
10. The QT interval (QTc) of 12-lead ECG is ≥450 ms for males and ≥470 ms for females.
11. There are risk factors that lead to prolonged QT interval or risk factors that increase arrhythmia, such as heart failure, ≥CTCAE (version 4.03) 2nd degree hypokalemia (2nd degree hypokalemia is defined as: serum potassium <the lower limit of the normal value is 3.0mmol/L, and there are symptoms and needs treatment), congenital long QT syndrome, family history of long QT syndrome.
12. Any drug known to prolong the QT interval is being used within 2 weeks before the first dose.
13. Insufficient bone marrow reserve or organ function, reaching any of the following laboratory limits (no corrective treatment within 1 week before laboratory examination of blood):

    1. Absolute neutrophil count <1.5×109 / L;
    2. Platelet count <90×109 / L;
    3. Hemoglobin <90 g/L (<9 g/dL);
    4. Alanine aminotransferase> 3 times the upper limit of normal (ULN);
    5. Aspartate aminotransferase>3×ULN
    6. Total bilirubin> 1.5×ULN;
    7. Creatinine> 1.5×ULN or creatinine clearance rate <45 mL/min (calculated by Cockcroft-Gault formula);
    8. Serum albumin (ALB) <28 g/L;
14. Female subjects who are pregnant, lactating, or planning to become pregnant during the study period.
15. A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of interstitial pneumonia requiring steroid therapy, or any evidence of clinically active interstitial lung disease.
16. Have a history of hypersensitivity to any active or inactive ingredients of Almonertinib, or to drugs with similar chemical structure to Almonertinib or in the same category as Almonertinib.
17. Any serious or uncontrolled eye disease (especially severe dry eye syndrome, dry keratoconjunctivitis, severe exposure keratitis or other diseases that may increase epithelial damage), according to the doctor's judgment, it may increase the safety risk of the subject; or patients with eye abnormalities who require surgery or are expected to require surgical treatment during the study period.
18. Use/consumption of drugs or foods that are known to have potent CYP3A4 inhibitory effects within 2 weeks, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefa Oxazolone, nelfinavir, ritonavir, saquinavir, telithromycin, aceto-eandomycin, voriconazole, and grapefruit or grapefruit juice.
19. Use drugs known to have potent CYP3A4 inducing effects within 2 weeks, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin and Hypericum perforatum.
20. Use drugs that are CYP3A4 substrates (with a narrow therapeutic index) within 2 weeks, including but not limited to dihydroergotamine, ergotamine, pimozide, astemizole, cisapride, and terfenadine.
21. Have used strong P-gp inhibitors (including but not limited to verapamil, cyclosporin A, dexverapamil) within 2 weeks.
22. Subjects judged by the investigator who may not be in compliance with the research procedures and requirements, such as subjects who have a clear history of neurological or mental disorders (including epilepsy or dementia), currently suffering from mental disorders, etc. .
23. The investigator judges that there are any subjects that endanger the safety of the subject or interfere with the evaluation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the anti-tumor activity by IRC: ORR | 8 weeks
  The objective response rate (ORR) was assessed by IRC for all eligible subjects after 8 weeks of Almonertinib induction therapy.
  Until the disease progresses or in the absence of disease progression, the last evaluable data will be recorded in the ORR assessment. However, any CR or PR that occurs after the termination of the study treatment and receiving further anti-tumor therapy will not be included in the ORR calculation.
Assess the anti-tumor activity by IRC: Event free survival (EFS) rate | 18 months
  The 18 months event-free survival period is defined as the time from random to the occurrence of any of the following events within 18 months, whichever occurs first:
  Tumor progression assessed by IRC according to RECIST 1.1; Tumor recurrence confirmed by IRC, including local recurrence or distant metastasis; Death caused by any cause.

SECONDARY OUTCOMES:
Assess the anti-tumor activity by investigators: ORR | 8 weeks
  The objective response rate (ORR) was assessed by investigators for all eligible subjects after 8 weeks of Almonertinib induction therapy.
  Until the disease progresses or in the absence of disease progression, the last evaluable data will be recorded in the ORR assessment. However, any CR or PR that occurs after the termination of the study treatment and receiving further anti-tumor therapy will not be included in the ORR calculation.
Assess the anti-tumor activity by investigators: Event free survival (EFS) | 18 months
  The 18 months event-free survival period is defined as the time from random to the occurrence of any of the following events within 18 months, whichever occurs first:
  Tumor progression assessed by investigators according to RECIST 1.1; Tumor recurrence confirmed by investigators, including local recurrence or distant metastasis; Death caused by any cause.
Event free survival (EFS) | 2 years
  The event-free survival period is defined as the time from random to the occurrence of any of the following events, whichever occurs first:
  Tumor progression assessed by IRC according to RECIST 1.1; Tumor recurrence confirmed by IRC, including local recurrence or distant metastasis; Death caused by any cause.
Overall survival (OS) | more than 2 years
  Overall survival is defined as the time between the date of first administration and the date of death of the subject for any reason.Subjects not dead at the time of the statistical analysis will be truncated at the time when the subject was last known to be alive.
Major pathological response (MPR) | 8 weeks
  The major pathological response rate is defined as the incidence of tumor regression induced by neoadjuvant therapy with pathological residual tumor ≤10% (only applicable to subjects who have received surgical treatment).
Assess the safety of Almonertinib | 2 years
  To evaluate number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Quality of life(QOL) assessed by EORTC QLQ-C30 | 2 years
  Quality of Life assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30(EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Kai can Cai, Principal Investigator — Nanfang Hospital, Southern Medical University; Guang Hai, Principal Investigator — Hubei Cancer Hospital; Hui Wang, Principal Investigator — Hunan Provincial Cancer Hospital; Hui Luo, Principal Investigator — Jiangxi Provincial Cancer Hospital; Qi xun Chen, Principal Investigator — Zhejiang Cancer Hospital; Dong Qian, Principal Investigator — Anhui Provincial Hospital; Zi li Meng, Principal Investigator — Huai 'an First People's Hospital; Di Ge, Principal Investigator — Shanghai Zhongshan Hospital; Yu sheng Su, Principal Investigator — Subei people's Hospital; Bao gang Liu, Principal Investigator — The Affiliated Cancer Hospital of Harbin Medical University; Yun peng Liu, Principal Investigator — First Hospital of China Medical University; Jun Zhao, Principal Investigator — Peking University Cancer Hospital & Institute; Qing song Pang, Principal Investigator — Tianjin Cancer Hospital; Bao sheng Li, Principal Investigator — Shandong Cancer Hospital and Institute; Yun chao Huang, Principal Investigator — Yunnan Cancer Hospital; Qi feng Wang, Principal Investigator — Sichuan Provincial Cancer Hospital; Ge Wang, Principal Investigator — Army Characteristic Medical Center of the People's Liberation Army; Jun Yao, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yan qiu Zhao, Principal Investigator — Henan Provincial People's Hospital; Wei hua Yang, Principal Investigator — Shanxi Provincial Cancer Hospital; Shuan ying Yang, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Guangdong Lung cancer institute, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No